CLINICAL TRIAL: NCT03328546
Title: Dietary Patterns and Health Outcomes (Cardiovascular, Metabolic, Endocrine, Neurological, Skeletal Muscular, Cancer)
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Walter C. Willett, NHS II Principal Investigator; Professor of Epidemiology and Nutrition, Harvard School of Public Health (HSPH)
Other Study IDs: NHS2/DPS-GEN; UM1CA176726 (NIH); K99ES026648 (NIH); K01DK103720-01 (NIH)
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Disorders; Metabolic Disease; Neoplasms; Endocrine System Diseases; Neurologic Symptoms; Skeletal Anomalies; Diabetes Mellitus; Pregnancy Complications
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders; Metabolic Diseases; Neoplasms; Endocrine System Diseases; Neurologic Manifestations; Diabetes Mellitus; Pregnancy Complications | interventions — Eating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dietary intake — Dietary intake converted into dietary pattern scores.

SUMMARY:
To study, prospectively, the association between dietary patterns and risk of health outcomes (cardiovascular, metabolic, endocrine, neurological, skeletal muscular, cancer) in cohort study of 116,671 women age 24 to 44 years at baseline in 1989 (the Nurses' Health Study II; NHS II).

DETAILED DESCRIPTION:
Health status and lifestyle information was self-reported on a questionnaire at baseline, and on questionnaires distributed to participants biennially thereafter. Dietary intake data was collected in form of a comprehensive, 131-item food frequency questionnaire (FFQ), distributed among participants every four years. The response rate remained over 90%. Dietary data was validated using biomarkers, health status data using medical records.

Dietary pattern scores were derived from FFQs using cumulative average whenever possible from years preceding the outcomes.

Multivariable Cox proportional hazards models were used to evaluate associations between dietary pattern scores and health outcomes, except in case of pregnancy complications (such as gestational diabetes mellitus/GDM and hypertensive disorders of pregnancy/HDPs) where multivariable logistic regression models with generalized estimating equations, with an exchangeable working correlation structure to account for correlated outcomes between pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* All women without history of chronic disease and/or primary outcome at the time of recruitment. Women contribute person-time until a first diagnosis of the primary outcome or until the end of follow-up.
* All women who reported a singleton pregnancy between 1991-2001 (data on pregnancy outcomes was collected on biennial questionnaires until 2001, since majority of women exited the reproductive age by then) (only for maternal outcomes)

Exclusion Criteria:

* women with a history of chronic disease (type 2 diabetes, cardiovascular disease, or cancer) or other disease studied as the primary outcome
* women with a missing or incomplete FFQ (more than 70 out of 131 items missing, or with caloric intake <800 kcal/day or >3500kcal/day) prior to endpoint.
* women with missing data on the primary outcome on biennial questionnaire.
* twin/multiple pregnancy (only for maternal outcomes)

Ages: 24 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Our analysis was based on a cohort of female registered nurses.
Study Population: The Nurses' Health Study II (NHS II) is a prospective cohort established in 1989 that includes 116,671 female registered U.S. nurses, aged 24-44 at baseline. Mailed questionnaires were administered biennially to collect data on medical and lifestyle factors, with a follow-up rate exceeding 90% for each 2-year cycle. Comprehensive food frequency questionnaires (FFQs) were distributed every four years to collect data on dietary intake.
Sampling Method: Non-Probability Sample
Enrollment: 116671 (Actual)
Dates: Start 1989-01-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction | 1989-2017
  Necrosis of heart muscle secondary to prolonged ischemia.
Coronary heart disease | 1989-2017
  Atherosclerosis
Stroke | 1989-2017
  Sudden death of brain cells due to lack of oxygen
Diabetes Mellitus (type 2) | 1989-2017
  Insulin resistance
Gestational Diabetes Mellitus | 1989-2017
  Glucose intolerance with onset/first recognition during pregnancy
Hypertensive disorders | 1989-2017
  Chronic hypertension
Hypertensive disorders of pregnancy | 1989-2001
  Pregnancy induced hypertension, toxemia/preeclampsia
Colon cancer | 1989-2017
  Malignant tumor in the colon
Breast cancer | 1989-2017
  Malignant tumor of breast cells
Fractures | 1989-2017
  Fragility fractures of common sites such as hip and wrist.
Physical functioning | 1989-2017
  Physical function such as falls, walking, and self care

CONTACTS AND LOCATIONS:
Overall Officials: Walter C. Willett, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)

IPD SHARING:
Plan to Share IPD: No
Data are de-identified

REFERENCES:
- [Background] Chiuve SE, Cook NR, Shay CM, Rexrode KM, Albert CM, Manson JE, Willett WC, Rimm EB. Lifestyle-based prediction model for the prevention of CVD: the Healthy Heart Score. J Am Heart Assoc. 2014 Nov 14;3(6):e000954. doi: 10.1161/JAHA.114.000954. PMID 25398889
- [Background] Chiuve SE, Fung TT, Rimm EB, Hu FB, McCullough ML, Wang M, Stampfer MJ, Willett WC. Alternative dietary indices both strongly predict risk of chronic disease. J Nutr. 2012 Jun;142(6):1009-18. doi: 10.3945/jn.111.157222. Epub 2012 Apr 18. PMID 22513989
- [Background] Bernstein AM, Pan A, Rexrode KM, Stampfer M, Hu FB, Mozaffarian D, Willett WC. Dietary protein sources and the risk of stroke in men and women. Stroke. 2012 Mar;43(3):637-44. doi: 10.1161/STROKEAHA.111.633404. Epub 2011 Dec 29. PMID 22207512
- [Result] Tobias DK, Zhang C, Chavarro J, Bowers K, Rich-Edwards J, Rosner B, Mozaffarian D, Hu FB. Prepregnancy adherence to dietary patterns and lower risk of gestational diabetes mellitus. Am J Clin Nutr. 2012 Aug;96(2):289-95. doi: 10.3945/ajcn.111.028266. Epub 2012 Jul 3. PMID 22760563
- [Result] Gaskins AJ, Rich-Edwards JW, Hauser R, Williams PL, Gillman MW, Penzias A, Missmer SA, Chavarro JE. Prepregnancy dietary patterns and risk of pregnancy loss. Am J Clin Nutr. 2014 Oct;100(4):1166-72. doi: 10.3945/ajcn.114.083634. Epub 2014 Aug 13. PMID 25240079
- [Result] Nimptsch K, Malik VS, Fung TT, Pischon T, Hu FB, Willett WC, Fuchs CS, Ogino S, Chan AT, Giovannucci E, Wu K. Dietary patterns during high school and risk of colorectal adenoma in a cohort of middle-aged women. Int J Cancer. 2014 May 15;134(10):2458-67. doi: 10.1002/ijc.28578. Epub 2013 Nov 25. PMID 24493161
- [Result] Malik VS, Fung TT, van Dam RM, Rimm EB, Rosner B, Hu FB. Dietary patterns during adolescence and risk of type 2 diabetes in middle-aged women. Diabetes Care. 2012 Jan;35(1):12-8. doi: 10.2337/dc11-0386. Epub 2011 Nov 10. PMID 22074723
- [Result] Willett WC, Stampfer MJ. Current evidence on healthy eating. Annu Rev Public Health. 2013;34:77-95. doi: 10.1146/annurev-publhealth-031811-124646. Epub 2013 Jan 7. PMID 23297654
- [Result] Schulze MB, Hoffmann K, Manson JE, Willett WC, Meigs JB, Weikert C, Heidemann C, Colditz GA, Hu FB. Dietary pattern, inflammation, and incidence of type 2 diabetes in women. Am J Clin Nutr. 2005 Sep;82(3):675-84; quiz 714-5. doi: 10.1093/ajcn.82.3.675. PMID 16155283
- [Result] Yu E, Rimm E, Qi L, Rexrode K, Albert CM, Sun Q, Willett WC, Hu FB, Manson JE. Diet, Lifestyle, Biomarkers, Genetic Factors, and Risk of Cardiovascular Disease in the Nurses' Health Studies. Am J Public Health. 2016 Sep;106(9):1616-23. doi: 10.2105/AJPH.2016.303316. Epub 2016 Jul 26. PMID 27459449